CLINICAL TRIAL: NCT00374517
Title: A Phase II Clinical Trial of Pimonidazole Hydrochloride as a Hypoxia Marker in Subjects Undergoing Elective Lung Resection for Treatment-Refractory Pulmonary Tuberculosis
Brief Title: Pimonidazole Hydrochloride to Detect Low Oxygen in Tuberculosis-Infected Lungs
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: International Tuberculosis Research Center (Other)
Responsible Party: Clifton E. Barry III, Ph.D./National Institute of Allergy and Infectious Diseases, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 999906241; 06-I-N241
Record Dates: First submitted 2006-09-08; First posted 2006-09-11 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-02-02

CONDITIONS: Refractory Pulmonary Tuberculosis
Keywords: Mycobacterium Tuberculosis; Pimonidazole Hydrochloride; Recurrent Tuberculosis; Hypoxyprobe; mRNA Expression; Pulmonary Tuberculosis
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis

INTERVENTIONS:
Drug: Pimonidazole hydrochloride

SUMMARY:
This study will determine whether a drug called pimonidazole hydrochloride shows areas of low oxygen in tuberculosis (TB)-infected lungs. Pimonidazole is a "low oxygen marker," an agent designed to find areas in the body that are not getting enough oxygen. If it is found that TB grows where oxygen is low, these results may help doctors decide what medicines would be most effective for treating TB.

Patients 20 years of age or older who are scheduled for lung surgery at the National Masan Tuberculosis Hospital in Masan, Korea to treat their TB may be eligible for this study.

Participants undergo the following procedures:

* Blood draw before surgery to test for hepatitis B and hepatitis C viruses.
* Pregnancy test for women who can become pregnant.
* Infusion of pimonidazole through a vein in the arm 24 hours before surgery. A part of the patient's lung is removed during surgery. This tissue is examined under a microscope for evidence of pimonidazole, which would indicate low oxygen.
* Blood sample collection during surgery and on the 7th and 14th days after surgery to check liver function.

DETAILED DESCRIPTION:
The purpose of this Phase II clinical trial is to establish whether pulmonary tuberculous lesions are hypoxic or contain hypoxic microenvironments using an in vivo hypoxia-imaging marker, pimonidazole hydrochloride, in subjects undergoing lung resection surgery for treatment-refractory pulmonary tuberculosis.

The study population will be drawn from subjects undergoing treatment at the National Masan Tuberculosis Hospital (NMTH), Masan, Republic of Korea. Subjects who are scheduled for partial lung resection surgery for treatment refractory TB will be eligible for this study. Selected subjects will be those who demonstrate one or more radiographic abnormalities associated with pulmonary tuberculosis (e.g., cavities, nodules, consolidation, fibrosis, or calcified lesions).

Subjects undergoing elective pulmonary resection will receive a single preoperative IV dose of pimonidazole 0.5 g/m(2) in 100 mL of normal saline, infused over 20 minutes 18 to 24 hours prior to surgery. The resected tissue will be analyzed to look at the following: 1) the degree of pimonidazole-adduct formation in tissue specimens with different histopathologic presentations; 2) the number of acid-fast bacilli in tissue sections, smears, or cultures prepared from homogenized lesions from distinct gross anatomic and histopathologic types in relation to the extent of tissue hypoxia, and; 3) comparison of lesions labeling with pimonidazole with the presence of human cellular and bacterial markers expected to be expressed under oxygen-limiting conditions. NIAID study investigators will have no input of any kind in selecting subjects for surgery, or in determining the kind or extent of surgical resection. Subjects will be on study from a few days before surgery until approximately 8 weeks after their surgery.

ELIGIBILITY:
* INCLUSION CRITERIA:

Males and females age 20 and above.

Subjects with treatment-refractory pulmonary TB (i.e., who remain sputum AFB smear positive and/or culture positive or who are sputum negative yet non-responsive by radiographic and clinical measures) (including MDR-TB) scheduled for elective pulmonary resection.

Subjects who demonstrate one or more radiographic abnormalities associated with pulmonary tuberculosis (i.e., cavities, nodules, consolidation, fibrosis, or calcified lesions).

Ability and willingness to utilize contraceptives (such as latex condom, diaphragm, cervical cap, IUD, hormonal contraception, tubal ligation, or vasectomy) from the time of consent to one month after the treatment period (both men and women).

Ability and willingness to give written or oral informed consent.

EXCLUSION CRITERIA:

Subjects under the age of 20.

Pregnant and breast-feeding women.

Subjects with underlying neurological disease including seizure disorder and peripheral neuropathy.

Subjects taking medications with a high incidence of central nervous system (CNS) toxicity (including cycloserine), within one week before or after the scheduled pimonidazole infusion or will be anticipated to need such drugs within one week after infusion.

Subjects taking the following medications within one week before or will be anticipated to need such drugs after the scheduled infusion: oral anticoagulants, Cimetadine, Didasnosine, Disulfiram, Nisatidine, Ocytetracycline, Phenobarbital, or Phenytoin.

Liver dysfunction with serum transaminases [AST (SGOT), ALT (SGPT)] and/or total bilirubin greater than 1.5 times ULN.

Evidence of hepatitis as indicated by a positive HBV surface antigen test or a positive HCV antibody titer suggesting chronic infection.

History of excessive alcohol use or alcohol abuse within the last year.

Renal insufficiency with serum creatinine greater than 1.5 times ULN.

Subjects assessed by the chest surgeon or surgery staff to be a high operative risk due to the presence of one or more underlying co-morbidities such as severe coronary artery disease, immunosuppression, or chronic obstructive pulmonary disease (COPD).

Administration of any investigational test article within 30 days preceding the first dose of study drug.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-09-05; Primary Completion 2010-02-02 (Actual); Study Completion 2010-02-02 (Estimated)

PRIMARY OUTCOMES:
Frequency of pimonidazole labeling in specific lesion types within resected lung specimens and the frequency of co-localization of AFB positive bacilli with pimonidazole regions in lesions. | Up to surgery.

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - International Tuberculosis Research Center, Masan
  - National Masan Tuberculosis Hospital, Masan

REFERENCES:
- [Background] Allen JG, Dische S, Lenox-Smith I, Malcolm SL, Saunders MI. The pharmacokinetics of a new radiosensitiser, Ro 03-8799 in humans. Eur J Clin Pharmacol. 1984;27(4):483-9. doi: 10.1007/BF00549599. PMID 6519157
- [Background] Durand RE, Raleigh JA. Identification of nonproliferating but viable hypoxic tumor cells in vivo. Cancer Res. 1998 Aug 15;58(16):3547-50. PMID 9721858
- [Background] Kennedy AS, Raleigh JA, Perez GM, Calkins DP, Thrall DE, Novotny DB, Varia MA. Proliferation and hypoxia in human squamous cell carcinoma of the cervix: first report of combined immunohistochemical assays. Int J Radiat Oncol Biol Phys. 1997 Mar 1;37(4):897-905. doi: 10.1016/s0360-3016(96)00539-1. PMID 9128967